CLINICAL TRIAL: NCT06988787
Title: Multifaceted Intervention to Restore Resilience and Overcome Risk
Acronym: MIRROR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Maria Kajankova, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 23-1671; HT94252410478 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Military Sexual Trauma; Intimate Partner Violence; Brain Injury; Post Traumatic Stress Disorder
Keywords: Military Sexual Trauma; Intimate Partner Violence; Female Veterans; Emotion Regulation; Brain Injury; Exposure Therapy
MeSH Terms: conditions — Military Sexual Trauma; Brain Injuries; Stress Disorders, Post-Traumatic; Emotional Regulation | interventions — Implosive Therapy

STUDY DESIGN:
Intervention Model Description: The proposed treatment study will employ a phase II RCT to evaluate whether the inclusion of an intervention that specifically targets EmReg (i.e., webSTAIR) prior to engaging in ExpoTx (webSTAIR+ ExpoTx) is more effective in improving outcomes/treatment effectiveness (PTSD symptomology and engagement) in FVets with MST and/or IPV and BI exposure. This treatment combination, (webSTAIR+ ExpoTx), will be compared to the standard EBP combination (PsychEd+ExpoTx). Participants will be randomized to one of the two intervention arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- webSTAIR+ExpoTx (Experimental): Web-based technology "webSTAIR" (Web-Based Skills Training in Affective Regulation and Interpersonal Relationships Program) will be used to guide Female Veterans (FVets) through each of the 10 webSTAIR skill modules for 5-weeks followed by 5 weeks of standard, patient-centered, exposure therapy (ExpoTx) delivered by a therapist.
  Interventions: Behavioral: webSTAIR; Behavioral: ExpoTx
- PsychoEd+ExpoTx (Active Comparator): 5 online sessions of psycho-education followed by 5 online sessions of exposure therapy
  Interventions: Behavioral: ExpoTx; Other: PsychoEd

INTERVENTIONS:
Behavioral: webSTAIR — Ten web-based modules that are completed independently by participants (~2 modules per week) and receive therapist support via video-telehealth after the completion of every 2 skill modules (1x per week for a total of 5 meetings).
  The first five modules review emotional awareness, emotion management, and distress tolerance while the final five modules raise awareness about relationship patterns and provide interpersonal skills training regarding effective assertiveness, interpersonal flexibility, and compassion for self and others.
  Other Names: Web-Based Skills Training in Affective Regulation and Interpersonal Relationships Program
  Arms: webSTAIR+ExpoTx
Behavioral: ExpoTx — A real-time, present-focused, intervention that does not require participants to relive or focus on past trauma(s), but rather on current social functioning; ie, how they are doing in day-to-day life, and current cognitive and psychological functioning. Therapist will meet individually with the participant for 5 sessions, 60 minutes each conducted virtually. During the 5 sessions, participants will be guided to use in vivo or in the moment ExpoTx to identified fear-based triggers. In each consecutive session, the therapist will engage the Veteran to explore cognitions that interfered with, reinforced, or diminished fear responses. Participants will be asked about their use of coping skills during exposure practice. Intentional participation in exposure for one target at least 30 minutes per day, or until SUDs lower by half. At the end of ExpoTx, the therapist will engage the Veteran in self-determining future goals and offer referrals in the community or at VA for additional support.
  Other Names: Exposure therapy
Other: PsychoEd — Psycho-education (PsychEd) orientation that provides an overview of PsychEd as a process for learning about mental health symptoms and disease management related to trauma. During PsychEd sessions, therapists will focus on the following 5 areas: 1) Defining trauma and PTSD. 2) Brain Basics and Brain Injury. 3) Understanding the Role of Stress and Its impact on trauma symptoms. 4) The Role of Nutrition and Exercise in Disease Management. 5) Information on other Programs.
  Other Names: Psycho-education
  Arms: PsychoEd+ExpoTx

SUMMARY:
The MIRROR study will compare the effectiveness of two interventions in improving emotion regulation and reducing PTSD symptoms in female Veterans with military sexual trauma (MST) and/or intimate partner violence (IPV) and co-occurring brain injury.

DETAILED DESCRIPTION:
Female Veterans (FVets) face disproportionately high rates of exposure to intimate partner violence (IPV) and military sexual trauma (MST). Studies suggest that a substantial proportion of women with MST and IPV exposure also experience co-occurring brain injury (BI) due to IPV/MST and from non-violent etiologies. Exposure to MST, IPV, and co-occurring BI, coupled with their effects on psychological outcomes, represents a significant health concern to both the military and public, yet there is a lack of effective interventions to treat the cumulative effects of MST, IPV and BI in FVets. The Multifaceted Intervention to Restore Resilience and Overcome Risk (MIRROR) study seeks to overcome this challenge by examining the effectiveness of a multifaceted intervention that combines a web-based emotion regulation (EmReg) intervention (Skills Training in Affective Regulation and Interpersonal Relationships program [webSTAIR]) and a Veteran's Affairs (VA) supported evidence-based practice (EBP), exposure therapy (ExpoTx), for treating post-traumatic stress disorder (PTSD) associated with MST, IPV, and BI in FVets. FVets who screen positive for exposure to MST and/or IPV, have a history of at least one BI, sub-threshold PTSD, and documented emotional dysregulation will be included and randomly assigned to either one of two intervention arms: 1) webSTAIR+ ExpoTx or 2) PsychEd+ ExpoTx. Aim 1 will examine the effectiveness of webSTAIR relative to psychoeducation (PsychEd) on EmReg in FVets with MST and/or IPV and BI. Aim 2 will examine whether improvements in EmReg lead to improved treatment outcomes in FVets. Aim 3 will examine the effectiveness of the interventions in maintaining treatment gains at the 3-month follow-up. The study will include lived experience consultants as research partners and involve a community advisory board (CAB) that includes FVets and key stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent as determined by UBACC, are English-speaking FVets who are 18+ years old
* Screen positive for exposure to IPV and/or MST using the VA Intimate Partner Violence Assistance Program (VA IPVAP) and MST Screening Protocol,
* Have a history of at least one BI assessed using the BISQ+IPV,
* Sub-threshold PTSD (operationalized as a total score of >33 on the PTSD Checklist Diagnostic and Statistical Manual of Mental Disorders-5 (PCL-5),
* Report deficits in Emotion Regulation (operationalized as a score of 0.5 SD above published means on the DERS).

Exclusion Criteria:

* FVets at high risk for suicide (respond yes to items 3, 4, 5, or 8 on the Columbia Suicide Severity Rating Scale [C-SSRS]),
* Observable active psychosis (e.g., auditory hallucinations, grandiose delusions),
* Those determined to have problematic substance use (score > 27 on the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) will be referred to substance use dependence programs for concurrent treatment. The PI and Co-Is will collaborate with the substance use dependence program to determine continued participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 136 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | At week 0, week 2.5, week 5, week 7.5, week 10, and month 3
  The DERS is a 36-item self-report measure that assesses emotion dysregulation in six domains: nonacceptance of emotional responses (subscale score 6-30), difficulties engaging in goal directed behavior (subscale score 5-25), impulse control difficulties (subscale score 6-30), lack of emotional awareness (subscale score 6-30), limited access to emotion regulation strategies (subscale score 8-40), and lack of emotional clarity (subscale score 5-25). Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Total Score range from 36-180, with higher scores indicating more difficulty in emotion regulation.

SECONDARY OUTCOMES:
Post-Traumatic Stress Disorder Checklist for the DSM-5 (PCL-5) | At week 0, week 2.5, week 5, week 7.5, week 10, and month 3
  The PCL-5 is a 20-item self-report measure that assesses DSM-5 criteria PTSD symptoms. Items are rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (extremely), and summed to compute the total scale that ranges from 0 to 80. Higher scores are indicative of greater symptom severity.
Depression and Anxiety Stress Scale (DASS) | At week 0, week 5, week 10, and month 3
  Depression Anxiety Stress Scales (DASS-42): A 42-item self-report measure assessing depression, anxiety, and stress. Each scale (14 items) is scored 0-3 per item, with total scores ranging 0-42 per domain. (Depression: Normal 0-9, Mild 10-13, Moderate 14-20, Severe 21-27, Extremely Severe 28+; Anxiety: Normal 0-7, Mild 8-9, Moderate 10-14, Severe 15-19, Extremely Severe 20+; Stress: Normal 0-14, Mild 15-18, Moderate 19-25, Severe 26-33, Extremely Severe 34+). Full scale from 0-126. Higher scores indicate greater severity.
Inventory of Interpersonal Problems (IIP-32) | At week 0, week 5, week 10, and month 3
  A 32-item measure used to screen for difficulties individuals experience in their interactions and relationships with others. The measure yields eight subscales of interpersonal problems including domineering/controlling, vindictive/self-centered, cold/distant, socially inhibited, nonassertive, overly accommodating, self-sacrificing, and intrusive/needy. Items are scored on a five-point scale from 0 (not at all) to 4 (extremely). Subscales ranges are 0-16, with full scale range 0-128, where higher score indicates greater intensity or frequency of interpersonal problems.
Dysexecutive Questionnaire (DEX) | At week 0, week 5, week 10, and month 3
  A 20-item self-report tool used to measure everyday problems associated with executive functioning difficulties. The DEX focuses on four domains: emotional, motivational, behavioral, and cognitive. Items are scored on a five-point scale from 0 (not at all) to 4 (extremely). Higher scores indicating greater reports of dysexecutive problems
Quality of Life after Brain Injury Overall Scale (QoLABRIOS) | At week 0, week 5, week 10, and month 3
  Six item self-report measure of global health related aspects of QoL after BI including physical condition, cognition, emotions, function in daily life, personal and social life, and current situation and future prospects. Full scale from 0-100, higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kajankova, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared, however, as required in study grant agreement, study team will upload a limited dataset to FITBIR.